CLINICAL TRIAL: NCT04723316
Title: Tumour Characterisation to Guide Experimental Targeted Therapy - National
Status: Recruiting | Type: Observational
Sponsor: The Christie NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CFTSp191
Record Dates: First submitted 2021-01-07; First posted 2021-01-25 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected for ctDNA analysis and germline DNA analysis Tissue samples will be collected for next generation sequencing. Whilst the focus of the study is on next generation sequencing of circulating tumour DNA, the study is not restricted to these analyses. Other tests may be performed, including, but not restricted to: immunohistochemistry, FISH, PCR if such analyses complement the panel of aberrations that may help select a relevant trial of an experimental therapeutic for participating patients.
  Fresh tumour may also be used for in vitro (i.e. organoids) and/or in vivo experiments (mouse models) (optional) if patients provide their consent. These crucial experiments will improve our understanding of the biology of cancer and will lead to identification of new potential targets for cancer patients, facilitate drug screening and will inform of mechanisms of drug resistance.
  In summary, analyses may be varied and alter over time as technologies evolve.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary aim of TARGET National is to establish a national framework to offer molecular profiling of circulating tumour DNA and/or tumour tissue (optional) to patients with advanced solid cancers referred to any of the Experimental Cancer Medicine Centres (ECMCs) across the UK, in order to help decision making for allocation to molecularly targeted experimental cancer treatments. Patients will be allocated treatment using a national Molecular Tumour Board to find the most suited therapies based on their molecular profiling results.

This study aims to recruit up to 6,000 patients with advanced solid tumours across 5 years and proposes to collect blood samples, archival tumour tissue and fresh tissue (optional)

The data may also be used for future development of predictive cancer biological markers, the design of clinical trials involving new or existing drugs, discovery of new genetic targets and exploring how resistance to specific anticancer agents arises in patients to help improve future cancer treatment management.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 16 years or over.
2. Written informed consent according to GCP and national regulations.
3. Patients with confirmed histological or cytological diagnosis of advanced solid cancer who have been referred to any of the ECMCs in the UK AND considered fit enough to receive an experimental therapeutic agent.
4. Availability of archival tumour sample (if tumour profiling is required)
5. Willingness to provide blood samples during the course of the study if allocated to a matched experimental therapy.

Exclusion Criteria:

1. Known HIV, Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or Hepatitis C virus (defined as HCV RNA detected), due to the difficulties in handling high-risk specimens. Routine testing for hepatitis is not required. Note: Patients with past/resolved Hepatitis B infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen [anti-HBc] antibody test) are eligible. Patients with a history of Hepatitis C infection are eligible only if polymerase chain reaction (PCR) analysis is negative for HCV RNA at least 6 months after completing treatment for Hepatitis C infection.
2. Known current COVID19 positive (by PCR) or active symptoms for COVID19. Routine testing for COVID19 is not required. Patients with past infection who have fully recovered may be included.
3. Patients who are unable to provide fully informed written consent.
4. Patients not considered eligible by the investigator for early phase clinical trials.
5. Patients currently receiving systemic anti-cancer therapy (due to potential impact on ctDNA analysis), unless patient has clear evidence of progression on hormone-based therapies or tyrosine kinase inhibitors. A minimum of 3 weeks is required post completion of other systemic anti-cancer therapies.
6. Presence of any medical, psychological, familial or sociological condition that, in the investigator's opinion, will hamper compliance with the study protocol and follow-up schedule.
7. Bleeding diathesis (patients' on anticoagulation are permitted to enter the trial if anticoagulation can be safely managed to enable fresh tumour biopsies and blood sampling).
8. Conditions in which research biopsies or blood sampling may increase risk of complications for the patients and/or investigator

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Potential study participants will be identified from patients with advanced solid cancer who have been referred for consideration of early phase clinical trials in ECMCs across the UK. Patients who meet the eligibility criteria and provide fully informed written consent will be enrolled into the study
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
To determine the number of patients matched to a trial of an experimental therapeutic agent based on molecular findings from ctDNA or tumour | 5 years

SECONDARY OUTCOMES:
Number of patients and cancer types with successful result obtained from ctDNA. | 5 years
Turnaround times from date of patient consent to date of genomic tumour profiling report generation. | 5 years
Number and range of molecular alterations found in blood (and/or tumour) of cancer patients referred to Experimental Cancer Medicine Centres. | 5 years
Overall response rates of patients who commence on a trial of an experimental therapeutic agent (matched or unmatched) on the basis of molecular findings in this study). | 5 years
Progression-free survival of patients who commence on a trial of an experimental therapeutic agent (matched or unmatched on the basis of molecular findings in this study). | 5 years
Overall survival of patients who commence on a trial of an experimental therapeutic agent (matched or unmatched on the basis of molecular findings in this study). | 5 years

CONTACTS AND LOCATIONS:
Locations (20):
- United Kingdom (20):
  - Queen's University Belfast, Belfast
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Cardiff University and Velindre Cancer Centre, Cardiff
  - Western General Hospital Edinburgh Cancer Centre, Edinburgh
  - Beatson West of Scotland Cancer Centre, Glasgow
  - St.James's University Hospital, Leeds
  - Leicester Cancer Research Centre, Leicester
  - Royal Free Hospital, London
  - Kings Health Partners, London
  - Imperial College London, London
  - UCL Cancer Institute, London
  - The Christie NHS Foundation Trust, Manchester
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Metropolitan Borough of Wirral
  - The Newcastle Upon Tyne NHS Foundation Trust, Newcastle
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - Royal Preston Hospital, Preston
  - Sheffield University Hospitals NHS Foundation Trust, Sheffield
  - University Hospitals Southampton NHS Foundation Trust, Southampton
  - ICR & The Royal Marsden, Sutton

IPD SHARING:
Plan to Share IPD: No